CLINICAL TRIAL: NCT04380857
Title: Assessing the Efficacy of DEXTENZA, Sustained Release Dexamethasone 0.4 mg Insert, When Placed Within the Lower Eye Lid Canaliculus in Comparison to Topical Prednisolone Acetate Following Bilateral Small Incision Lenticule Extraction (SMILE)
Brief Title: Assessing Dextenza Insert After SMILE Procedure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: William Wiley, MD (Other)
Responsible Party: Sponsor-Investigator, William Wiley, MD, Principal Investigator, Cleveland Eye Clinic
Organization: Cleveland Eye Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WW-2020-DexSMILE
Record Dates: First submitted 2020-05-05; First posted 2020-05-08 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Post Procedural Infection
MeSH Terms: interventions — Calcium Dobesilate; prednisolone acetate

STUDY DESIGN:
Intervention Model Description: First eye randomized for either topical prednisolone acetate (control eye) or lower eyelid canaliculus Dextenza insertion (study eye) and the contralateral eye receiving opposite treatment in the OR following SMILE
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexamethasone ophthalmic insert 0.4 mg (Experimental): Dexamethasone ophthalmic insert 0.4 mg
  Interventions: Drug: Dexamethasone ophthalmic insert 0.4 mg
- Topical prednisolone acetate ophthalmic drops (Active Comparator): topical prednisolone acetate ophthalmic drops
  Interventions: Drug: Topical Prednisolone Acetate Ophthalmic Drops

INTERVENTIONS:
Drug: Dexamethasone ophthalmic insert 0.4 mg — intracanalicular dexamethasone insert
  Other Names: Dextenza
  Arms: Dexamethasone ophthalmic insert 0.4 mg
Drug: Topical Prednisolone Acetate Ophthalmic Drops — Topical Prednisolone acetate ophthalmic drops per standard of care:
  Every two hours on day of procedure, then four times a day for the first week, then two times a day for the second week, then discontinue
  Other Names: Prednisolone Acetate
  Arms: Topical prednisolone acetate ophthalmic drops

SUMMARY:
This three-month prospective, open-label, single-center, randomized investigator initiated clinical study seeks to investigate the efficacy of DEXTENZA when placed in the lower canaliculus (study eye) compared to topical corticosteroids (control eye) following bilateral SMILE surgery. In addition, the study will evaluate physician assessment of ease of DEXTENZA insertion

DETAILED DESCRIPTION:
4.1 Study Population The study aims to enroll 20 patients undergoing bilateral SMILE.

4.1.1 Inclusion Criteria

A patient's study eye must meet the following criteria to be eligible for inclusion in the study:

* Age 18 years and older
* Scheduled for bilateral SMILE surgery
* Willing and able to comply with clinic visits and study related procedures
* Willing and able to sign the informed consent form

4.1.2 Exclusion Criteria

A patient who meets any of the following criteria will be excluded from the study:

* Patients under the age of 18.
* Pregnancy (must be ruled out in women of child-bearing age with pregnancy test)
* Active infectious systemic disease
* Active infectious ocular or extraocular disease
* Obstructed nasolacrimal duct in the study eye(s)
* Hypersensitivity to dexamethasone
* Patients being treated with immunomodulating agents in the study eye(s)
* Patients being treated with immunosuppressants and/or oral steroids Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Scheduled for bilateral SMILE surgery
* Willing and able to comply with clinic visits and study related procedures
* Willing and able to sign the informed consent form

Exclusion Criteria:

* Patients under the age of 18.
* Pregnancy (must be ruled out in women of child-bearing age with pregnancy test)
* Active infectious systemic disease
* Active infectious ocular or extraocular disease
* Obstructed nasolacrimal duct in the study eye(s)
* Hypersensitivity to dexamethasone
* Patients being treated with immunomodulating agents in the study eye(s)
* Patients being treated with immunosuppressants and/or oral steroids Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Wiley, MD, Principal Investigator — Cleveland Eye Clinic
Locations (1):
- Cleveland Eye Clinic, Brecksville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective, randomized, fellow-eye controlled study was conducted at a single site (Clear Choice Custom LASIK Center) in 20 patients (40 eyes) with three surgeons between June 2020 and June 2021 and was performed according to guidelines established by the Declaration of Helsinki.
Pre-assignment Details: Twenty-three patients were enrolled in the study. One patient failed screening and was not randomized. Two additional patients were randomized, but the Dextenza insert could not be successfully placed in the assigned eye at the time of surgery.
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Dexamethasone Ophthalmic Insert 0.4 mg | Topical Prednisolone Acetate Ophthalmic Drops
Started | 20; 20 Eyes | 20; 20 Eyes
Completed | 17; 17 Eyes | 17; 17 Eyes
Not Completed | 3; 3 Eyes | 3; 3 Eyes
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Enrolled Patients: Enrolled patients who underwent SMILE surgery in both eyes with investigational treatment in one eye and standard of care treatment in the fellow eye.
Arm/Group | Enrolled Patients
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Pain
Description: post-op pain as measured as scores on an Ocular Pain Assessment Scale from 0-10 ("0" being no pain and "10" being the worst pain you could imagine)
Time Frame: Change is being assessed at Baseline, Day 1, Day 7, Day 30 and Day 90
Population: All subjects were seen through week 1; three were lost to follow up thereafter.
Measure: Mean (Standard Deviation); unit: Score on a scale from 0-10
Units Other Than Participants: Eyes
Arm/Group | Dexamethasone Ophthalmic Insert 0.4 mg | Topical Prednisolone Acetate Ophthalmic Drops
Number analyzed (Participants) | 20 | 20
Number analyzed (Eyes) | 20 | 20
Score on a scale from 0-10
  Pre-operative | 0.15 (0.5) | 0.20 (0.5)
  Day 1 | 0.95 (1.36) | 0.90 (1.12)
  Day 7 | 0.47 (0.94) | 0.37 (0.67)
  Day 30: number analyzed (Participants) | 17 | 17
  Day 30: number analyzed (Eyes) | 17 | 17
  Day 30 | 0.41 (1.7) | 0.06 (0.24)
  Day 90: number analyzed (Participants) | 17 | 17
  Day 90: number analyzed (Eyes) | 17 | 17
  Day 90 | 0 (0) | 0 (0)

2. Secondary Outcome: Number of Lines Lost From Best Corrected Visual Acuity
Description: After manifest refraction all units assessed for best corrected distance visual acuity using ETDRS. Number of lines seen was then converted to LogMar score (on a scale of -0.30 to 1.00 where smaller numbers indicate better vision and larger numbers indicate worse vision) to measure changes in Best Corrected Distance Visual Acuity between Baseline and Day 90
Time Frame: Baseline through Day 90
Population: All subjects were seen through week 1; three were lost to follow up thereafter.
Measure: Mean (Full Range); unit: Score on a scale
Units Other Than Participants: Eyes
Arm/Group | Dexamethasone Ophthalmic Insert 0.4 mg | Topical Prednisolone Acetate Ophthalmic Drops
Number analyzed (Participants) | 17 | 17
Number analyzed (Eyes) | 17 | 17
Score on a scale | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Loss of Lines in Uncorrected Visual Acuity
Description: All units assessed for uncorrected visual acuity using ETDRS. Number of lines seen was then converted to LogMar to measure changes in uncorrected visual acuity between Baseline and Day 90.
Time Frame: Baseline to Day 7, Day 30 and Day 90
Population: All subjects were seen through week 1; three were lost to follow up thereafter.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Dexamethasone Ophthalmic Insert 0.4 mg | Topical Prednisolone Acetate Ophthalmic Drops
Number analyzed (Participants) | 20 | 20
Number analyzed (Eyes) | 20 | 20
logMAR
  1 week | -0.010 (0.0114) | 0.013 (0.183)
  1 month: number analyzed (Participants) | 17 | 17
  1 month: number analyzed (Eyes) | 17 | 17
  1 month | -0.014 (0.181) | -0.026 (0.160)
  3 months: number analyzed (Participants) | 17 | 17
  3 months: number analyzed (Eyes) | 17 | 17
  3 months | -0.071 (0.108) | -0.068 (0.156)

4. Secondary Outcome: Post op Pain Management Per Eye
Description: Count of participants requiring pain management from Day 0 to Day 90.
Time Frame: Day 0 to Day 90
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Dexamethasone Ophthalmic Insert 0.4 mg | Topical Prednisolone Acetate Ophthalmic Drops
Number analyzed (Participants) | 17 | 17
Number analyzed (Eyes) | 17 | 17
Eyes | 0 | 0

5. Secondary Outcome: Patient Preference Between Groups
Description: As reported by patients choosing one of five options; Strongly preferred insert, preferred insert, no preference, preferred standard drop regimen, strongly preferred standard drop regimen.
Time Frame: Day 7, Day 30 and Day 90
Population: All subjects were seen through week 1; three were lost to follow up thereafter.
Measure: Count of Participants; unit: Participants
Groups:
- No Preference: No Preference
Arm/Group | Dexamethasone Ophthalmic Insert 0.4 mg | Topical Prednisolone Acetate Ophthalmic Drops | No Preference
Number analyzed (Participants) | 20 | 20 | 20
Participants
  Day 7 | 14 | 2 | 4
  Day 30: number analyzed (Participants) | 17 | 17 | 17
  Day 30 | 11 | 3 | 3
  Day 90: number analyzed (Participants) | 17 | 17 | 17
  Day 90 | 9 | 3 | 5

ADVERSE EVENTS:
Time Frame: Baseline to 90 Days
Arm/Group | Dexamethasone Ophthalmic Insert 0.4 mg | Topical Prednisolone Acetate Ophthalmic Drops
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone Ophthalmic Insert 0.4 mg (N=20) | Topical Prednisolone Acetate Ophthalmic Drops (N=20)
Intraocular pressure elevation (Eye disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT04380857/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT04380857/SAP_002.pdf